CLINICAL TRIAL: NCT00053157
Title: Use Of Granulocyte Macrophage Colony Stimulating Factor (GM-CSF) To Mobilize Donor Peripheral Blood Stem Cells Along With GM-CSF Administration Post Allogeneic Transplant - A Pilot Study
Brief Title: Sargramostim in Reducing Graft-Versus-Host Disease in Patients Who Are Undergoing Donor Stem Cell Transplantation for Hematologic Cancer or Aplastic Anemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Purpose: Supportive Care
Other Study IDs: RPC 02-01; RPCI-RPC-0201
Record Dates: First submitted 2003-01-27; First posted 2003-01-28 (Estimated); Last update posted 2022-10-05 (Actual); Status verified 2022-10

CONDITIONS: Chronic Myeloproliferative Disorders; Graft Versus Host Disease; Leukemia; Lymphoma; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasms
Keywords: graft versus host disease; accelerated phase chronic myelogenous leukemia; chronic phase chronic myelogenous leukemia; primary myelofibrosis; childhood acute myeloid leukemia/other myeloid malignancies; childhood acute promyelocytic leukemia (M3); recurrent childhood acute lymphoblastic leukemia; recurrent childhood acute myeloid leukemia; recurrent childhood large cell lymphoma; recurrent childhood lymphoblastic lymphoma; recurrent childhood small noncleaved cell lymphoma; recurrent/refractory childhood Hodgkin lymphoma; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; meningeal chronic myelogenous leukemia; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II mantle cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult Burkitt lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult acute lymphoblastic leukemia; recurrent adult acute myeloid leukemia; recurrent adult Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; relapsing chronic myelogenous leukemia; secondary acute myeloid leukemia; refractory chronic lymphocytic leukemia; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult Burkitt lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage III chronic lymphocytic leukemia; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult Burkitt lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; stage IV chronic lymphocytic leukemia; untreated adult acute lymphoblastic leukemia; untreated adult acute myeloid leukemia; untreated childhood acute lymphoblastic leukemia; untreated childhood acute myeloid leukemia and other myeloid malignancies; childhood chronic myelogenous leukemia; chronic eosinophilic leukemia; chronic neutrophilic leukemia; atypical chronic myeloid leukemia, BCR-ABL1 negative; myelodysplastic/myeloproliferative neoplasm, unclassifiable; noncontiguous stage II small lymphocytic lymphoma; noncontiguous stage II marginal zone lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with t(15;17)(q22;q12); childhood myelodysplastic syndromes
MeSH Terms: conditions — Myeloproliferative Disorders; Graft vs Host Disease; Leukemia; Lymphoma; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Leukemia, Myeloid, Accelerated Phase; Leukemia, Myeloid, Chronic-Phase; Primary Myelofibrosis; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Dendritic Cell Sarcoma, Interdigitating; Burkitt Lymphoma; Recurrence; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Leukemia, Myeloid, Acute; Hodgkin Disease; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Leukemia, Lymphocytic, Chronic, B-Cell; Pdgfra-Associated Chronic Eosinophilic Leukemia; Leukemia, Neutrophilic, Chronic; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Lymphoma, B-Cell, Marginal Zone; Congenital Abnormalities | interventions — sargramostim

INTERVENTIONS:
Biological: sargramostim

SUMMARY:
RATIONALE: Colony-stimulating factors such as sargramostim may increase the number of immune cells found in bone marrow or peripheral blood and may help a person's immune system recover from the side effects of chemotherapy or radiation therapy. Giving sargramostim to the stem cell donor and the patient may reduce the chance of developing graft-versus-host disease following stem cell transplantation.

PURPOSE: Clinical trial to study the effectiveness of sargramostim in decreasing graft-versus-host disease in patients who are undergoing donor stem cell transplantation for hematologic cancer or aplastic anemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of sargramostim (GM-CSF) to mobilize CD34+ hematopoietic stem cells in donors and to reduce graft-vs-host disease in patients after allogeneic stem cell transplantation (SCT) for hematologic malignancy or aplastic anemia.
* Determine the safety of GM-CSF after allogeneic SCT transplantation in these patients.

OUTLINE: This is a pilot study.

* Donors: Donors receive sargramostim (GM-CSF) subcutaneously (SC) once daily on days 1-6. Donors undergo stem cell harvest on day 7.

Donors may undergo up to 3 apheresis procedures to reach the target stem cell dose and may receive additional GM-CSF prior to each collection.

* Patients: Patients receive conditioning therapy as per transplantation protocol RP98-15. Patients undergo allogeneic stem cell transplantation on day 0. Patients then receive GM-CSF SC once daily beginning on day 7 and continuing until blood counts recover.

Patients are followed weekly until day 100 and then at days 180 and 360.

PROJECTED ACCRUAL: A total of 10 patients and 10 donors will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of a malignant hematologic disease, including:

  * Acute or chronic leukemia
  * Myelodysplastic syndromes
  * Myeloproliferative disorder
  * Hodgkin's lymphoma
  * Non-Hodgkin's lymphoma OR
* Aplastic anemia
* Planned transplantation on an RPCI IRB-approved allogeneic stem cell transplantation protocol
* HLA-matched (6/6) related donor available

PATIENT CHARACTERISTICS:

Age

* 5 to 60

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients and donors must use effective contraception
* No known allergy to GM-CSF
* No prior of adverse reaction to any yeast recombinant molecule

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics
* No prior allogeneic stem cell transplantation

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Ages: 5 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2002-06; Primary Completion 2004-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip L. McCarthy, MD, Study Chair — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States